CLINICAL TRIAL: NCT00067210
Title: Cooling of the Head and Neck to Reduce Seizure Frequency: A Pilot Study
Brief Title: Reducing Seizure Frequency Using Cooling of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Susumu Sato, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030272; 03-N-0272
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-13

CONDITIONS: Epilepsy; Seizures
Keywords: Brain; Epilepsy; Core; Temperature
MeSH Terms: conditions — Epilepsy; Seizures

INTERVENTIONS:
Device: Head and Neck Cooling System

SUMMARY:
Doctors use cooling of the brain to help stop seizures. This procedure is usually accomplished through surgery. Cooling of the face and scalp may also cool the brain, avoiding the need for surgery.

The purpose of this study is to assess a head-neck cooling device that the patient can wear. Researchers will determine whether the device can change the frequency of seizures in people with epilepsy.

Study participants must be 21 years of age or older and must experience seizures that occur once a week on a regular basis. Participants will be asked to keep a detailed seizure diary for a 12-week period before the date of the first cooling session. For each of the four cooling sessions, participants will be admitted to the hospital overnight. They will undergo a physical and neurological exam and an EEG (electroencephalogram). They will also swallow a temperature-sensor pill. Participants will have one 60-minute cooling session once a week for 4 weeks. Investigators will paste temperature-sensing electrodes on the scalp, forearm, abdomen, and leg. Participants will then be fitted with the cooling unit and the session will begin.

DETAILED DESCRIPTION:
Previous experimental as well as clinical reports have clearly shown that cooling of the brain does have inhibitory effects on epileptiform discharges and seizures. We hypothesize that mild cooling of the brain has anti-epileptic effects in epileptic patients who either have no identifiable seizure foci, who have multiple foci, or who have frequent localization-related seizures that are refractory to antiepileptic drugs. We have studied the feasibility and safety of a head-neck cooling device in 10 adult normal volunteers, and found that the head-neck cooling was feasible and safe, without significant complaints or problems voiced by the subjects. Overall, a slight reduction of core temperature was shown. Since cooling on a twice-a-week basis was well tolerated by normal volunteers, we would like to extend our study to patients with epilepsy to learn the optimal duration and frequency of head-neck cooling in terms of reducing seizure frequency. This will be a pilot study, as directed by PIRC and the IRB, in which we will evaluate 60 minutes of cooling performed once a week for 4 weeks in 5 epileptic patients. We will then report the results to PIRC and the IRB before we proceed with further study.

ELIGIBILITY:
* INCLUSION CRITERIA:

A minimum of one documented seizure of any type per a 1-week period.

21 years or older, and able to cooperate with the cooling procedures.

On a stable antiepileptic drug (AED) regimen, as determined by history and by AED plasma levels as measured in the CC OPD.

The ability to maintain a daily seizure calendar, either independently or with help from a family member.

No history of intestinal problems or history of intestinal surgery.

Must be able to swallow medication in capsule form.

EXCLUSION CRITERIA:

Female patients who are pregnant.

Those patients under 21 years of age.

Those patients who may have difficulty swallowing a large capsule, or describing their feelings and experiences related to the cooling sessions.

Those patients with a history of intestinal problems or intestinal surgery

Those patients with progressive neurological disorders

Those sensitive to coldness

History of severe 'ice-cream' headache

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2003-08-11; Study Completion 2007-05-22

PRIMARY OUTCOMES:
Identify optimal cooling parameters,namely duration and frequency of cooling for reducing seizure frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cabanac M. Selective brain cooling in humans: "fancy" or fact? FASEB J. 1993 Sep;7(12):1143-6; discussion 1146-7. doi: 10.1096/fasebj.7.12.8375612.